CLINICAL TRIAL: NCT01015248
Title: Multicentric, Non-Randomized Phase 2 Trial of Bendamustine And Rituximab for Patients With Previously Untreated Extranodal Mucosa-Associated Lymphoid Tissue (MALT) Lymphoma
Brief Title: Trial of Bendamustine And Rituximab for Patients With Previously Untreated Extranodal Mucosa-Associated Lymphoid Tissue (MALT) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MALT2008-01; No EudraCT: 2008-007725-39
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: MALT LYMPHOMA
Keywords: CD 20 positive
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab and Bendamustine (Experimental)
  Interventions: Drug: Rituximab and Bendamustine

INTERVENTIONS:
Drug: Rituximab and Bendamustine — Rituximab 375 mg/m2 iv. day 1 Bendamustine 90 mg/m2 iv. day 1 and 2

SUMMARY:
The aim of the study is to assess the therapeutic activity and safety of the combination of Bendamustine and Rituximab in MALT lymphomas.

Primary endpoint:

* Event-free-survival (EFS) (failure or death from any cause) for all patients.

Secondary endpoints:

* Complete and partial remission rates for all patients
* Response duration (time to relapse or progression) for responder patients
* Progression-free-survival (PFS) (disease progression or death from lymphoma: for all patients
* Overall survival for all patients
* Acute and long-term toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of CD20-positive marginal zone B-cell lymphoma of MALT type arisen at any extranodal site (WHO classification)
2. Any stage (Ann Arbor I-IV)
3. The novo disease en any extranodal site. For primary gastric or cutaneous lymphoma, local/specific previous treatment is accepted, just following the below criteria:

   1. Cutaneous lymphoma: recurrent lymphoma after local therapy
   2. Gastric lymphoma:

   b1. H. pylori-negative cases, either de novo (non pre-treated) or at relapse following local therapy (i.e., surgery, radiotherapy or antibiotics).

   b2. H. pylori-positive cases at diagnosis, who failed antibiotic therapy, including patients with: clinical (endoscopic) and histological evidence of disease progression at any time post H. pylori eradication; stable disease with persistent lymphoma at 1 year post H. pylori eradication; relapse (without H. pylori re-infection), after a remission; patients who failed either first line antibiotics or further local treatment (surgery or radiotherapy)
4. No evidence of histologic transformation to a high grade lymphoma
5. Measurable or evaluable disease
6. Age >18 and <85
7. ECOG performance status 0-2
8. Life expectancy of at least 1 year
9. Written informed consent given according to national/local regulations

Exclusion Criteria:

1. Prior chemotherapy or prior immunotherapy with any anti-CD20 monoclonal antibody
2. Prior radiotherapy in the last 6 weeks
3. Corticosteroids during the last 28 days, unless prednisone chronically administered at a dose <20 mg/day for indications other than lymphoma or lymphoma-related symptoms
4. Major impairment of renal function (serum creatinine > 2,5 x upper normal) or liver function (ASAT/ALAT <2,5 x upper normal, total bilirubin <2,5x upper normal), unless due to lymphoma involvement.
5. Impairment of bone marrow function (WBC <3.0x109/L, ANC <1.5x109/L, PLT <100x109/L), unless due to lymphoma involvement
6. Evidence of clinically significant cardiac, neurological or metabolic disease, unless due to lymphoma involvement
7. Evidence of symptomatic central nervous system (CNS) disease
8. Active HBV and/or HCV infection
9. Known HIV infection
10. Prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer
11. Any psychiatric disease potentially hampering compliance with the study protocol and follow-up schedule
12. Potential to attend regular visits to the hospital, on an outpatient regimen
13. Hypersensibility to any compound of the study medication.
14. Non appropriate contraceptive method in women of childbearing potential or men
15. Treatment with any drug under research within 30 days previous to start the study medication.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of assessment is the event-free-survival (EFS) according to the criteria of the International Workshop to Standardize Response Criteria for NHL and Criteria for evaluation of response in NHL | 2 years follow-up

SECONDARY OUTCOMES:
Include evaluation of the next parameters: Complete and partial remission rates for all patients Response duration for responder patients PFS for all patients Overall survival for all patients Acute and long-term toxicity | 2 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Montalbán, MD, Principal Investigator — Ramon y Cajal Hospital; Antonio Salar, MD, Principal Investigator — Hospital del Mar; Ana Muntañola, MD, Principal Investigator — Mutua de Terrassa Hospital; Mª José Rodríguez, MD, Principal Investigator — Hospital Universitario de Canarias; María José Terol, MD, Principal Investigator — Hospital Clínico de Valencia; Juan Manuel Sancho, MD, Principal Investigator — ICO Hospital Germans Trias i Pujol; Eva Domingo, MD, Principal Investigator — ICO Hospital Durans i Reynals; Grande Carlos, MD, Principal Investigator — 12 de Octubre Hospital; Carlos Panizo, MD, Principal Investigator — Clínica Universitaria Navarra; Miguel Canales, MD, Principal Investigator — La Paz Hospital; Raquel Oña, MD, Principal Investigator — MD Anderson Hospital; Reyes Arranz, MD, Principal Investigator — La Princesa Hospital; Dolores Caballero, MD, Principal Investigator — Hospital Unisversitario de Salamanca; José Luis Bello, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago; Joan Bargay, MD, Principal Investigator — Son Llátzer Hospital; Luis Palomera, MD, Principal Investigator — Hospital Clínico de Zaragoza; Franciaco Javier Peñalver, MD, Principal Investigator — Fundación Hospital Alcorcón; Eulogio Conde, MD, Principal Investigator — Marqués de Valdecilla Hospital; José Javier Sánchez-Blanco, MD, Principal Investigator — Morales Meseguer Hospital; Concepción Nicolás, MD, Principal Investigator — Central de Asturias Hospital
Locations (19):
- Spain (19):
  - ICO-Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - ICO-Hospital Durans i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Fundación Alcorcón, Alcorcón, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital MD Anderson, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Son Llátzer, Palma de Mallorca, Mallorca
  - Hospital Morales Meseguer, Murcia, Murcia
  - Clínica Universitaria Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital Clínico de Zaragoza "Lozano Blesa", Zaragoza, Zaragoza

REFERENCES:
- [Derived] Salar A, Domingo-Domenech E, Panizo C, Nicolas C, Bargay J, Muntanola A, Canales M, Bello JL, Sancho JM, Tomas JF, Rodriguez MJ, Penalver FJ, Grande C, Sanchez-Blanco JJ, Palomera L, Arranz R, Conde E, Garcia M, Garcia JF, Caballero D, Montalban C; Grupo Espanol de Linfomas/Trasplante de Medula Osea (GELTAMO). First-line response-adapted treatment with the combination of bendamustine and rituximab in patients with mucosa-associated lymphoid tissue lymphoma (MALT2008-01): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2014 Dec;1(3):e104-11. doi: 10.1016/S2352-3026(14)00021-0. Epub 2014 Nov 19. PMID 27029228